CLINICAL TRIAL: NCT01926730
Title: Food and Crohn's Exacerbation Study (FACES)
Acronym: FACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K24-DK078228-FACES; K24DK078228 (NIH)
Record Dates: First submitted 2013-08-18; First posted 2013-08-21 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual diet (No Intervention): Patients will follow a usual diet and consume at least 16 oz of water per day
- Restriction diet (Experimental): Participants will follow a diet that limits intake of selected food items. Patients will consume at least 16 oz of water per day.
  Interventions: Other: Restriction diet

INTERVENTIONS:
Other: Restriction diet — Selected food items will be limited in the participants diet
  Arms: Restriction diet

SUMMARY:
The proposed study is a randomized controlled trial of a limited restriction diet compared to a regular diet among patients with Crohn's disease (CD) in remission. At baseline, patients will complete a semi-quantitative food frequency questionnaire assessing usual dietary patterns over the preceding month. Disease activity will be assessed with the abbreviated Crohn's Disease Activity Index (aCDAI)59. Self-reported disease status will be assessed during follow-up using an internet-based questionnaire. Repeat assessment of adherence to the study diets will be assessed with food frequency questionnaires (FFQs) administered after 20 weeks. Follow-up duration will be for 48 weeks. Statistical analysis will compare the time to relapse using Cox regression for patients in the two study arms. In the exploratory aim, we will compare outcomes among patients in the highest tertile for other food items and nutrients to those in the lowest tertile based on self-reported usual dietary patterns at baseline. Thus, the study population will be analyzed both as a randomized controlled trial and as a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an established diagnosis of CD.
2. All patients must be in clinical remission at the time of entry into the study. Remission is defined as an aCDAI of less than 150.

Exclusion Criteria:

Inflammatory bowel disease (IBD) unspecified / Indeterminate colitis

Total or sub-total colectomy, ileostomy, or colostomy

Unable to read and speak English

No internet access

Steroids other than budesonide ≤6mg/day with the prior two weeks

Perianal fistula or abscess with more than scant drainage

Age less than 18 years

Pregnant or breastfeeding women

Unwilling to follow the study diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Relapse of Crohn's Disease (CD) | Every 8 weeks during the 48 week study period
  Relapse of CD is defined as an increase in the aCDAI by >=60 points and to >150. Additionally, undergoing CD surgery or starting any new CD medication (steroids, mesalamine, azathioprine, methotrexate, anti-Tumor Necrosis Factor α (anti-TNF), anti-α4) for the treatment of CD symptoms during the interval between two visits will be considered to have identified a clinical relapse.

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States